CLINICAL TRIAL: NCT01629927
Title: Evaluation of Phenotypic and Genetic Properties in Male Subjects Affected By Hypohidrotic Ectodermal Dysplasia (ECP-012)
Acronym: ECP-012
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-012
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: X-linked Hypohidrotic Ectodermal Dysplasia; Hypohidrotic Ectodermal Dysplasia
Keywords: X-linked hypohidrotic ectodermal dysplasia; Hypohidrotic ectodermal dysplasia; HED; XLHED
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HED-affected males: Male subjects affected by HED
- Male controls: Male subjects not affected by HED

SUMMARY:
The study proposes to enroll male subjects affected by Hypohidrotic Ectodermal Dysplasia (XLHED). The sweat duct images will be acquired with a CE marked skin-imaging device and the sweat rate will be measured using a CE marked pilocarpine iontophoresis and collection system. The technologies for both imaging of sweat ducts and the measurement of maximal sweat rate have been used safely and without adverse events in our prior studies involving HED/XLHED subjects. Furthermore, this study will assess the feasibility of developing a non-invasive screening tool that will enable detection of clinical signs of XLHED based on an analysis of a two dimensional frontal photograph.

DETAILED DESCRIPTION:
The study proposes to enroll male subjects affected by XLHED (determined by genetic testing and restricted to age > 1 yr). The sweat duct images will be acquired with a CE marked skin-imaging device and the sweat rate will be measured using a CE marked pilocarpine iontophoresis and collection system. The technologies for both imaging of sweat ducts and the measurement of maximal sweat rate have been used safely and without adverse events in our prior studies involving HED/XLHED subjects. Furthermore, this study will assess the feasibility of developing a non-invasive screening tool that will enable detection of clinical signs of XLHED based on an analysis of a two dimensional frontal photograph.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled in this study.

* Attending the 2012 Spanish Association for those Affected by Ectodermal Dysplasia Annual Reunion;
* One year of age or greater;
* Conform to one of the following requirements for providing informed consent/assent:

  * If more than 18 years of age, subjects must provide signed informed consent;
  * If less than 18 years of age and it is determined that the subject is capable of providing assent, both the assent of the subject and consent of the parent(s) or guardian of that subject must be granted. Under this condition, both parents of the subject should give their permission, unless 1 parent is deceased, unknown, incompetent, or not available;
  * If the subject is incapable of providing assent, the consent of the parent(s) or guardian of the subject must be granted. Under this condition, both parents should give their consent, unless 1 parent is deceased, unknown, incompetent, or not available.
* Can provide documentation of genetic testing results positive for an EDA gene mutation /deletion;
* As described in Section 3.2 above, subjects must meet one of the following criteria:

  * Documented diagnosis of XLHED confirmed via genetic testing;
  * Unaffected male controls.

Exclusion Criteria:

* Known hypersensitivity to pilocarpine or pilocarpine-like muscarinic agonists;
* Presence of pacemakers;
* Subjects who are not able or are not willing to comply with the procedures of this protocol;
* Subjects with any major medical problem that will prevent them from participating in this study.

Min Age: 1 Year | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study is being conducted among family members attending the 2012 Spanish Association for those Affected by Ectodermal Dysplasia Annual Reunion, March 30-April 1, 2012, at the Center for Rare Diseases in Burgos, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Collecting demographic and clinical status information in XLHED affected males and unaffected male siblings using a medical questionnaire and clinical photographs | Study day 1 - Day of study conduct
Assess the feasibility of developing a non-invasive newborn screening tool, which will enable detection of clinical symptoms of HED/XLHED at birth, based on an analysis of a two dimensional photograph | Study day 1 - Day of study conduct

SECONDARY OUTCOMES:
The secondary objective of this descriptive study is to use skin assessment techniques to characterize skin properties in male subjects affected by XLHED compared with unaffected male sibling controls, including determination of the number of sweat ducts | Study day 1 - Day of study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Encarna Navarro, MD, PhD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Center for Rare Diseases, Burgos, Spain